CLINICAL TRIAL: NCT00817167
Title: Open Label, Randomized, Comparative, Single Center, Pilot Study to Assess the Added Value of inReach Technology Software on Performance Characteristics of Standard Bronchoscopy.
Brief Title: Added Value of inReach Software on Performance Characteristics of Standard Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: superDimension Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DPR0006
Record Dates: First submitted 2009-01-01; First posted 2009-01-06 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Lung Disease
Keywords: Known or suspected lung disease; Candidates for non-emergency bronchoscopy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- inReach (A) (Experimental): Bronchoscopy procedure is planned using inReach planning software
  Interventions: Device: inReach bronchoscopy planning software
- Control (B) (Active Comparator): Bronchoscopy procedure is planned using standard CT viewer software
  Interventions: Device: Standard lung CT viewer

INTERVENTIONS:
Device: inReach bronchoscopy planning software — inReach planning software creates three-dimensional lung CT reconstruction, enabling rapid virtual endoscopic depiction of the airways that allows to plan bronchoscopy virtually.
  Arms: inReach (A)
Device: Standard lung CT viewer — CT viewer, used for standard bronchoscopy
  Arms: Control (B)

SUMMARY:
The study is aimed to evaluate and describe the added value of inReach planning software on performance characteristics of standard bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for non-emergency bronchoscopy
* Must provide signed informed consent
* Male or female above 18 years old
* Lung lesions up to 3 cm in size (in largest diameter), non-visible by standard bronchoscope

Exclusion Criteria:

* CT done over a month before the bronchoscopy procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Bronchoscopy Diagnostic Yield, compared between two study groups and calculated as percentage of true diagnoses from total number of bronchoscopy procedures. | Until the definitive diagnosis is obtained

SECONDARY OUTCOMES:
Bronchoscopy Safety Profile, compared between two groups and calculated as percentage of bronchoscopy-related adverse events. | At discharge from bronchoscopy unit

CONTACTS AND LOCATIONS:
Overall Officials: Avi Mann, MD, Principal Investigator — Pulmonology Department, Tel Aviv Sourasky Medical Center
Locations (1):
- Pulmonology Department, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Schwarz Y, Greif J, Becker HD, Ernst A, Mehta A. Real-time electromagnetic navigation bronchoscopy to peripheral lung lesions using overlaid CT images: the first human study. Chest. 2006 Apr;129(4):988-94. doi: 10.1378/chest.129.4.988. PMID 16608948
- [Background] Gildea TR, Mazzone PJ, Karnak D, Meziane M, Mehta AC. Electromagnetic navigation diagnostic bronchoscopy: a prospective study. Am J Respir Crit Care Med. 2006 Nov 1;174(9):982-9. doi: 10.1164/rccm.200603-344OC. Epub 2006 Jul 27. PMID 16873767
- [Background] Eberhardt R, Anantham D, Herth F, Feller-Kopman D, Ernst A. Electromagnetic navigation diagnostic bronchoscopy in peripheral lung lesions. Chest. 2007 Jun;131(6):1800-5. doi: 10.1378/chest.06-3016. Epub 2007 Mar 30. PMID 17400670
- See also: superDimension Inc. — http://www.superdimension.com